CLINICAL TRIAL: NCT00332891
Title: An 8-Week, Double-Blind, Placebo-Controlled, Multicenter Study With Paroxetine (20 mg q24) as Positive Control, Evaluating the Efficacy and Safety of 2 Fixed Doses of SR58611A (175 mg q12 and 350 mg q12) in Outpatients With GAD
Brief Title: An Eight-Week Study to Evaluate the Efficacy and Safety of SR58611A in Patients With Generalized Anxiety Disorder
Acronym: ELECTRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5891
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety Disorders
Keywords: Anxiety; Anti-Anxiety Agents; controlled Clinical Trials
MeSH Terms: conditions — Anxiety Disorders | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SR58611A in patients with Generalized Anxiety Disorder. The primary objective is to evaluate the efficacy of a 350 mg and 700 mg dose of SR58611A compared to placebo in patients with generalized anxiety disorder (GAD). The secondary objectives are to evaluate the efficacy of SR58611A on disability and quality of life in patients with GAD and to evaluate safety of SR58611A

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from generalized anxiety disorder (GAD) as defined by DSM-IV-TR criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) plus GAD Module
* Total score on the 14-item Hamilton Anxiety Rating Scale (HAM-A) equal or above 20.

Exclusion Criteria:

* Patients with a diagnosis of Major Depressive Disorder as defined by DSM-IV-TR within 6 months of study entry.
* Patients with a Montgomery-Asberg Depression Rating Scale (MADRS) total score of 18 or higher at screening or baseline visits.
* Patients having a moderate to high current risk for suicide.
* Patients with other current anxiety disorder assessed with the MINI: agoraphobia, social phobia, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, acute stress disorder.
* Patients with a lifetime history according to the MINI of: bipolar disorders, psychotic disorders, antisocial personality disorder.
* Patients with severe or unstable concomitant medical conditions according to the Investigator's judgment.
* Females who are pregnant or lactating.
* Female patients of childbearing potential must use an effective method of birth control during the entire study period.
* Patients with positive test for any illicit drug included in the urine drug screen.
* Participation in a clinical trial of an experimental therapy within 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2006-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the change from baseline to Day 56 of treatment in the Hamilton Anxiety Rating Scale (HAM-A) total score.

SECONDARY OUTCOMES:
The main secondary outcomes are the changes from baseline to Day 56 of treatment in the CGI Severity of Illness Score, percentage of patients with HAM-A treatment response and change from baseline in the HAM-A somatic and psychic anxiety factor scores.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Belgrade, Serbia

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com